CLINICAL TRIAL: NCT05884320
Title: Phase II Trial of Sacituzumab Govitecan in Recurrent and/or Metastatic Secretory Gland Cancers
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0813; NCI-2023-04260 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-05-22; First posted 2023-06-01 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Gland; Salivary Gland Cancers
MeSH Terms: conditions — Salivary Gland Neoplasms | interventions — sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1: ACC (Experimental): Paritcipants will receive sacituzumab govitecan by vein on Days 1 and 8 of each cycle. The first dose will be given over about 3 hours. All other doses will be given over about 1-2 hours. Premedication for prevention of infusion reactions will be administered prior to each sacituzumab govitecan infusion.
  Interventions: Drug: Sacituzumab Govitecan
- Cohort 2: Non-ACC (Experimental): Paritcipants will receive sacituzumab govitecan by vein on Days 1 and 8 of each cycle. The first dose will be given over about 3 hours. All other doses will be given over about 1-2 hours. Premedication for prevention of infusion reactions will be administered prior to each sacituzumab govitecan infusion.
  Interventions: Drug: Sacituzumab Govitecan

INTERVENTIONS:
Drug: Sacituzumab Govitecan — Given by IV (vein)

SUMMARY:
To learn if sacituzumab govitecan can help to control salivary gland cancer.

DETAILED DESCRIPTION:
Primary Objectives:

* To assess the efficacy of SG in patients with R/M secretory gland carcinomas, specifically ACC (cohort 1) and SDC, adeno-NOS, and MEC (cohort 2)

Secondary Objectives:

* To estimate the median duration of response (DOR)
* To estimate the median progression-free survival (PFS)
* To estimate the median overall survival (OS)
* To assess safety of SG

Tertiary / Exploratory Objectives:

* To explore biomarkers that may predict response to therapy

ELIGIBILITY:
Inclusion Criteria:

All patients must meet all of the following inclusion criteria to be eligible for participation in this study:

1. Patients ≥18 years with histology-proven R/M salivary gland cancer.
2. Not amenable to curative intent surgery or radiotherapy
3. Measurable disease per RECIST 1.1
4. Performance status ECOG of 0 or 1
5. Patient has provided informed consent.
6. Laboratory measurements, blood counts:

   1. Hemoglobin ≥ 9 g/dL. Red blood cell transfusions are permitted to meet the hemoglobin inclusion criteria
   2. Absolute neutrophil count ≥ 1 x 10^9/mL without growth factor support for 28 days
   3. Platelets ≥ 100 x 10^9/mL without platelet transfusion for 28 days
7. Laboratory measurements, renal function:

   Creatinine clearance ≥ 30 mL/min as assessed by the Cockcroft-Gault equation
8. Laboratory measurements, hepatic function:

   1. AST and ALT ≤ 2.5 x ULN or ≤ 5 x ULN in patients with liver metastases
   2. Total bilirubin ≤ 1.5 x ULN or ≤ 3.0 x ULN and primarily unconjugated if patient has a documented history of Gilbert's syndrome or genetic equivalent
9. Female patients with reproductive potential must practice two effective contraceptive measures for the duration of study drug therapy and for at least 90 days after completion of study therapy. The two birth control methods can be either two barrier methods or a barrier method plus a hormonal method to prevent pregnancy. The following are considered adequate barrier methods of contraception: diaphragm, condom, copper intrauterine device, sponge, or spermicide. Appropriate hormonal contraceptives will include any registered and marketed contraceptive agent that contains an estrogen and/or a progesterone agent (including oral, subcutaneous, intrauterine, or intramuscular agents).
10. Male patients who are sexually active with women with reproductive potential must agree to use contraception for the duration of treatment and for at least 90 days after completion of study therapy.

    Cohort 1:

    In addition to meeting the inclusion criteria for all patients, patients who are enrolled into Cohort 1 must fulfill the following cohort-specific inclusion criteria:
11. Patients with histology-proven R/M ACC who are treatment-naïve or received any number of prior systemic therapy in the setting of R/M disease.
12. Disease progression per RECIST within 6 months or unequivocal clinical progression within 6 months per investigator's assessment.

    Cohort 2:

    In addition to meeting the inclusion criteria for all patients, patients who are enrolled into Cohort 2 must fulfill the following cohort-specific inclusion criterion:
13. 13) Patients with histology-proven R/M SDC or intermediate or high-grade adenocarcinoma NOS, or intermediate or high grade MEC, who progressed on up to 3 lines of palliative chemotherapy in the R/M setting. Any number of prior targeted-therapy, hormonal therapy, and/or immunotherapy are allowed.
14. Patients with HER2 overexpressing (3+ by IHC) or amplified tumors, must have received at least one prior line with a HER2-targeting agent OR must have a contra-indication for HER-2 targeted therapy (Eg: reduced left ventricular ejection fraction).

Exclusion Criteria:

Patients who meet any of the following exclusion criteria are not eligible to be enrolled in this study:

1. Prior radiation therapy (or other non-systemic therapy) within 2 weeks prior to enrollment
2. Active CNS disease (patients with asymptomatic and stable, treated CNS lesions who have been off corticosteroids, radiation, or other CNS-directed therapy for at least 4 weeks are not considered active)
3. Red blood cell transfusion dependence, defined as requiring more than 2 units of packed RBC transfusions during the 4-week period prior to screening. Red blood cell transfusions are permitted during the screening period and prior to enrollment to meet the hemoglobin inclusion criterion.
4. Prior anticancer therapy including, but not limited to, chemotherapy, immunotherapy, or investigational agents within 4 weeks or 5 half-lives prior to SG treatment
5. Current participation in another interventional clinical study
6. History of previous malignancy other than malignancy treated with curative intent. Patients with the following diagnoses represents an exception and may enroll if ≥ 1 year with no evidence of active disease before the first dose of the study drug.:

   1. Non-melanoma skin cancers with no current evidence of disease
   2. Melanoma in situ with no current evidence of disease
   3. Localized cancer of the prostate with prostate-specific antigen of <1 ng/mL
   4. Treated or localized well-differentiated thyroid cancer
   5. Treated cervical carcinoma in situ
   6. Treated ductal/lobular carcinoma in situ of the breast
7. Evidence of uncontrolled, active infection, requiring systemic anti-bacterial, anti-viral or anti-fungal therapy ≤ 10 days prior to administration of investigational product. Patients with known hepatitis B, hepatitis C (HCV), or HIV infection could go on study provided the viral load is undetectable at screening.
8. Disease or medical conditions that would substantially increase the risk-benefit ratio of participating in the study that include: acute myocardial infarction within the last 6 months, unstable angina, uncontrolled diabetes mellitus, significant active infections, and congestive heart failure New York Heart Association Class III-IV
9. Female patients who are pregnant or breast-feeding
10. Known hypersensitivity to any of the study drugs, the metabolites, or formulation excipient
11. Received a live-virus vaccination within 30 days of planned treatment start. Seasonal flu vaccines that do not contain live virus are permitted.
12. High dose systemic corticosteroids (≥ 20 mg of prednisone or its equivalent) are not allowed within 2 weeks of study treatment (C1D1).
13. Cognitively impaired patients who are incompetent to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-27 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Renata Ferrarotto, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Siqueira JM, Mitani Y, Marques-Piubelli ML, Hoff CO, Bonini F, de Sousa LG, Mitani M, Carvalho GL, Nunes FD, Matos LL, Lin SY, Spiotto MT, Hanna EY, McGrail DJ, El-Naggar AK, Ferrarotto R. TROP2 Expression in Salivary Gland Adenoid Cystic Carcinoma (ACC) According to Histologic Subtype: Therapeutic Implications. J Oral Pathol Med. 2025 Sep;54(8):658-666. doi: 10.1111/jop.70008. Epub 2025 Jul 8. PMID 40624990
- See also: M D Anderson Cancer Center — http://www.mdanderson.org